CLINICAL TRIAL: NCT06898840
Title: Study to Examine Glycaemic Responses to the Ingestion of Fruit Juices and Smoothies Using Different Measurement Methodologies.
Brief Title: Establishing the Glycaemic Index of Fruit Drinks Using Different Measurement Methodologies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Emma Greatorex Brooks, PhD Researcher, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 7134-9931
Record Dates: First submitted 2025-02-28; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-01

CONDITIONS: Glycaemic Index; Glycaemic Response Measurements
Keywords: Fruit Drinks; Glycaemic Index

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, replicate crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- CONTROL (Active Comparator): 50 g glucose (55 g dextrose powder accounting for hydration) plus 641 mL water
  Interventions: Other: Fruit drink
- REPLICATE CONTROL (Active Comparator): 50 g glucose (55 g dextrose powder accounting for hydration) plus 641 mL water
  Interventions: Other: Fruit drink
- S&B (Experimental): 417 mL of commercially available "Strawberries & Bananas" fruit smoothie providing 50 g carbohydrate [strawberries (31%), apples, bananas (22%), white grapes, oranges, blackcurrants]. Plus 224 mL water to standardise volume
  Interventions: Other: Fruit drink
- REPLICATE S&B (Experimental): 417 mL of commercially available "Strawberries & Bananas" fruit smoothie providing 50 g carbohydrate [strawberries (31%), apples, bananas (22%), white grapes, oranges, blackcurrants]. Plus 224 mL water to standardise volume
  Interventions: Other: Fruit drink
- OJ (Experimental): 641 mL of commercially available "Smooth Orange Juice" providing 50 g of carbohydrate [100% oranges]
  Interventions: Other: Fruit drink
- AJ (Experimental): 455 mL commercially available "Apple Juice" providing 50 g of carbohydrate [apples, ascorbic acid]. Plus 186 mL water to standardise volume
  Interventions: Other: Fruit drink
- ENERGISE (Experimental): 417 mL of commercially available "Energise Super Smoothie" providing 50 g carbohydrate [apples (50%), red grapes, bananas, strawberries (10%), blackcurrants, sour cherries (3.3%), pressed beetroot, flax seeds (0.56%), guarana infusion (0.01%), vitamins B1, B2, B3, B6, C & E]. Plus 224 mL water to standardise volume
  Interventions: Other: Fruit drink
- BLUE (Experimental): 521 mL of commercially available "Bolt from the Blue" juice drink providing 50 g carbohydrate [apple (66%), coconut water (18%), white grapes, white guava (5.2%), passion fruit, lime (0.87%), spirulina extract (0.81%) vitamins B1, B2, B3, B6, C & E]. Plus 120 mL water to standardise volume
  Interventions: Other: Fruit drink

INTERVENTIONS:
Other: Fruit drink — Commercially available fruit drinks or smoothies

SUMMARY:
Glycaemic responses to carbohydrates ingested as fruit sugars may vary depending on factors inherent to the fruit and the type of sugar. The aim of this project is to investigate the glycaemic responses to a range of commercially available fruit drinks and to establish the glycaemic index for each product relative to a glucose reference. Differences in recorded responses could also be influenced by the sample type (capillary blood vs interstitial fluid) and participant characteristics. Participants will ingest 8 test drinks including 5 different fruit drinks (OJ, AJ, S&B, ENERGISE, BLUE), each matched for carbohydrate to the glucose reference (CONTROL) which will be sampled two times, an additional sample of one of the smoothies (S&B) will also be replicated. Fingerstick capillary blood sampling alongside dual sited continuous glucose monitors (CGM) will measure glucose and lactate concentrations, subjective appetite sensations will also be recorded. The tests will follow best practice guidelines for glycaemic index testing. These data will provide insight into how differing formulations can alter the glycaemic responses to fruit drinks, and whether sampling technique can affect the interpretations of measurement.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Body mass index 18-30 kg/m2

Exclusion Criteria:

* diagnosis of any form of diabetes
* intolerances or allergies to any of the study procedures (e.g. fructose/inulin intolerance)
* Fructose malabsorption
* Inborn errors of fructose metabolism (e.g. fructokinase deficiency, aldolase B deficiency, fructose-1,6-bisphosphatase deficiency)
* pregnant or lactating
* any condition that could introduce bias to the study (e.g. diagnoses of lipid disorders, including cardiovascular disease, or therapies that alter lipid or glucose metabolism, such as statins or niacin).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Glycaemic indices for 5 test drinks measured using capillary blood samples | 120 minutes
  Glycaemic indices [2-hour incremental area under the glucose curve (mmol/L-1x120 minutes) for each of the 5 test drinks relative to mean value of control conditions (CONTROL, REPLICATE CONTROL), expressed as a percentage] in capillary blood samples

SECONDARY OUTCOMES:
Glycaemic index of all conditions with capillary blood samples vs CGM | 120 minutes
  The difference in glycaemic index [2-hour incremental area under the glucose curve (mmol/L-1x120 minutes) for 5 test drinks relative to mean control (CONTROL, REPLICATE CONTROL), expressed as a percentage] in capillary blood samples versus continuous glucose monitors.

OTHER OUTCOMES:
Comparisons between conditions in glucose concentration in capillary samples | 120 minutes
  Comparison of blood glucose concentration 2-hour incremental area under the curve (iAUC) min.mmol/L between test conditions
Comparisons between conditions in glucose concentration in capillary samples | 120 minutes
  Comparison of postprandial peak concentration mmol/L of blood glucose between test conditions (Cmax)
Comparisons between conditions in glucose concentration in capillary samples | 120 minutes
  Comparison of time to peak blood glucose concentration in minutes (Tmax) between test conditions
Comparisons between conditions in glucose concentration in capillary samples | 120 minutes
  Comparison of blood glucose concentration mmol/L at 2 hours between test conditions
Comparisons between conditions in glucose concentration with CGM | 120 minutes
  Comparison of glucose concentration 2-hour incremental area under the curve (iAUC) min.mmol/L between test conditions
Comparisons between conditions in glucose concentration with CGM | 120 minutes
  Comparison of postprandial peak concentration mmol/L of glucose between test conditions (Cmax)
Comparisons between conditions in glucose concentration with CGM | 120 minutes
  Comparison of time to peak glucose concentration in minutes (Tmax) between test conditions
Comparisons between conditions in glucose concentration with CGM | 120 minutes
  Comparison of glucose concentration mmol/L at 2 hours between test conditions
Comparisons between conditions in lactate concentration in capillary samples | 120 minutes
  Comparison of blood lactate concentration 2-hour incremental area under the curve (iAUC) min.mmol/L between test conditions
Comparisons between conditions in lactate concentration in capillary samples | 120 minutes
  Comparison of postprandial peak concentration mmol/L of blood lactate between test conditions (Cmax)
Comparisons between conditions in lactate concentration in capillary samples | 120 minutes
  Comparison of time to peak blood lactate concentration in minutes (Tmax) between test conditions
Comparisons between conditions in lactate concentration in capillary samples | 120 minutes
  Comparison of blood lactate concentration mmol/L at 2 hours between test conditions
Comparisons between conditions of appetite ratings | 120 minutes
  Comparison of subjective appetite sensations assessed with visual analogue scales (2-hour area under the curve min.mmVAS)
Comparisons between individuals | 120 minutes
  Comparison of Postprandial lactate concentration min.mmol/L between individuals 2-hour incremental area under curve (iAUC)
Comparisons between individuals | 120 minutes
  Comparison of Postprandial glucose concentration min.mmol/L between individuals 2-hour incremental area under curve (iAUC)
Comparisons between individuals | 120 minutes
  Comparison of Appetite rating responses min.mmVAS between individuals 2-hour area under curve (AUC)
Comparisons within individuals | 120 minutes
  Comparison within individuals of interstitial glucose concentrations measurements from continuous glucose monitors on left and right arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available open access on the University of Bath Research Data Archive (RDA) at the point of publication in a peer-reviewed journal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: These will become available at the point of publication permanently
URL: https://researchdata.bath.ac.uk/

REFERENCES:
- [Background] Gonzalez JT. Are all sugars equal? Role of the food source in physiological responses to sugars with an emphasis on fruit and fruit juice. Eur J Nutr. 2024 Aug;63(5):1435-1451. doi: 10.1007/s00394-024-03365-3. Epub 2024 Mar 16. PMID 38492022